CLINICAL TRIAL: NCT04165551
Title: A Double-blind, Randomized, Controlled, Parallel Groups Study for the Evaluation of the Effects of the Consumption of Lactobacillus BSL_PS71 on the Load of Streptococcus Agalactiae on Vaginal Mucosa.
Brief Title: Evaluation of the Consumption of a Probiotic on the Load of S. Agalactiae.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosearch S.A. (Industry)
Collaborators: Federico García García, PhD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P048
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-08

CONDITIONS: Streptococcus Agalactiae
Keywords: Streptococcus agalactiae; ProbioticsPrevention
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Volunteers will take 1 capsule per day containing 6x109 cfu of Lactobacillus BSL_PS71 in maltodextrin.
  Interventions: Biological: Probiotic
- Placebo (Placebo Comparator): Volunteers will take 1 capsule per day containing maltodextrin.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Probiotic — Volunteers will take 1 capsule a day of the Probiotic during lunch without any restrictions on diet or lifestyle.
  Arms: Probiotic
Biological: Placebo — Volunteers will take 1 capsule a day of the Placebo during lunch without any restrictions on diet or lifestyle.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effects of oral administration of Lactobacillus BSL_PS71 on the presence of S. agalactiae in vaginal microbiota of healthy women.

DETAILED DESCRIPTION:
Group B streptococci (Streptococcus agalactiae) are found in the vaginal microbiota in 10-30% of women without showing signs of infection. However, during delivery, it can be transmitted to the baby and, although in most cases it does not lead to disease, in a percentage of 5% of babies it causes serious infections that can trigger the death of the baby. In order to avoid this risk, a protocol of intra-partum preventive administration of antibiotics was implanted decades ago in women with a positive vaginal culture for this species in the weeks before birth. Taking into account the high percentage of women who show positive culture, this represents a high percentage of women who receive preventive antibiotic treatment with the consequences that this has for the mother's and baby's microbiota, as well as contributing to the generation of antibiotic resistance, a serious problem for today's society.

The fecal microbiota is considered a source of bacteria for the vaginal microbiota. In fact, women who present S. agalactiae in the vaginal microbiota also have it in stool. Given the demonstrated ability of Lactobacillus to control certain bacterial populations, the ability of a battery of Lactobacillus strains to inhibit the growth of S. agalactiae in the context of the fecal microbiota was analyzed. From these tests the strain Lactobacillus BSL_PS71 was selected for its antibacterial capacity against S. agalactiae.

ELIGIBILITY:
Inclusion Criteria:

* Test positive for S. agalactiae in vaginal exudate
* Accept freely to participate in the study and sign the informed consent document

Exclusion Criteria:

* Consumption of probiotic supplements
* Antibiotic use in the period of 2 weeks before the start of the study
* Being pregnant or intending to get pregnant in the next 8 weeks
* Being allergic to any group of antibiotics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
Detection of Streptococus agalactiae in vaginal exudate | 8 weeks
  It will be determined the presence of S. agalactiae in vaginal exudate

SECONDARY OUTCOMES:
Cuantification of bacterial populations in vaginal exudate | 8 weeks
  It will be cuantified the bacterial populations in vaginal exudate

CONTACTS AND LOCATIONS:
Overall Officials: Federico García, PhD, Study Chair — Head of the Microbiology Service at the San Cecilio Hospital (Granada, Spain)
Locations (1):
- Biosearch Life, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No